CLINICAL TRIAL: NCT04787796
Title: The Application of a Portable Multichannel ECG System for the Patients Suspected to Have Possible Coronary Artery Disease or Acute Coronary Syndromes
Brief Title: The Application of a Portable Multichannel ECG System for the Patients Suspected to Have Possible CAD or ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201905108DIND
Record Dates: First submitted 2020-05-19; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2020-05

CONDITIONS: CAD
Keywords: CAD，ACS，Multichannel ECG recorder
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Self-built-in M-ECG recorders have passed the electrical. (Experimental): We shall conduct this prospective clinical study to define the specific patterns of multichannel ECG change in adults with suspected CAD or ACS. For multichannel ECG (M-ECG) examination, the signal will be recorded with a Self-built-in ECG recorder.
  Interventions: Device: a 28-channel ECG (MECG) system

INTERVENTIONS:
Device: a 28-channel ECG (MECG) system — To test if a 28-channel ECG (MECG) system would efficiently differentiate the patients suspected to have CAD or ACS with acceptable sensitivity and specificity, and optimize this portable self-built-in multichannel ECG recorder system with various algorithms.

SUMMARY:
This clinical trial is to test if a 28-channel ECG (MECG) system would efficiently differentiate the patients suspected to have CAD or ACS with acceptable sensitivity and specificity, and optimize this portable self-built-in multichannel ECG recorder system with various algorithms. The 28-channel ECG (MECG) system is a multi-channel real-time cardiovascular performance evaluation system. The system mainly includes: a multi-channel ECG signals measurement unit, a multi-channel ECG signals processing device, and an ECG signals reconstruction unit. The method uses a MAMA-END algorithm, to mark ECG signals to replace the original ECG signal and to extract and reconstruct a first signals having QRS wave, and a second signal having T wave; then method detects and marks the start of Q wave and the end of T wave on the first signal and the second signal. Therefore, the method is able to determine and evaluate if a patient does have cardiovascular disease, and to locate the lesion positions of a patient having cardiovascular disease.

DETAILED DESCRIPTION:
We shall conduct this prospective clinical study to define the specific patterns of multichannel ECG change in adults with suspected CAD or ACS. For multichannel ECG (M-ECG) examination, the signal will be recorded with a Self-built-in ECG recorder. However, the examinations, diagnosis, medications, or procedures for the patients will only depend on the decision made by the primary care physicians through the traditional ways. The M-ECG results will not be used by the primary physicians for any diagnosis or decision-making of the patients. That is, the final diagnosis of CAD will be made with coronary angiography and the final diagnosis of ACS will be made with the traditional criteria (symptoms, traditional ECG changes, and cardiac enzyme changes).

Multichannel ECG Study The Self-built-in M-ECG recorders have passed the electrical security test. Multichannel ECG study will be performed under the approval of the Institutional Review Board. Before ECG examination, subjects will receive adequate orientation of the examination procedures and will complete inform consent.

During the ECG recording ,the patent will lie down flat on the bed, and 4 ECG leads with commercially available pads (Covidien Kendall ECG electrodes Medi-trace 200) will be applied on the 4 extremities, respectively. Using xyphoid process as a right lower reference point, a 18cm x 18cm patch integrated with 24 evenly distributed electrode pads (Covidien Kendall ECG electrodes Medi-trace Mini 100) will be applied on the left chest wall . Then, the ECG signals will be recorded through the self-built-in ECG recorders. The overall period for recording will be around 10 minutes.

The postprocessing and analysis of the ECG data will be performed with a PC computer by an analyzer without prior knowledge of the patient's clinical information. After ECG data is acquired, the analytic software will provide an electrical mapping of QTc dispersion (SIQTC).

ELIGIBILITY:
Inclusion Criteria:

1. >20 years
2. Patients admitted for cardiac catheterization examination due to clinically suspected coronary artery disease (CAD): Those who have exertional chest pain and positive ischemic change by stress test, highly suspected lesions on non-invasive images, or very typical chest pain symptoms.
3. Patients visiting ER due to suspected ACS: Those who have sudden onset of chest pain or shortness of breath.

Exclusion Criteria:

1. Wound over the fore chest
2. Life-threatening malignancy in 5 years
3. Treatment with immunosuppressive agents
4. Any unfeasible condition or situation from the opinion of the primary care physicians (ex.

critical condition needing emergency treatment or intervention, cardio pulmonary cerebral resuscitation, etc.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The existence of coronary stenosis on coronary angiogram | 3 days
  ECG QTc dispersion > 72 msec on Multichannel ECG

SECONDARY OUTCOMES:
Localization of myocardial ischemia | 3 days
  Channel numbers of ECG QTc < 400 msec on Multichannel ECG

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Tien Chang, Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No